CLINICAL TRIAL: NCT02429531
Title: The Polysaccharide Antibody Response Study: Typhim Vi Response and Allohemagglutinins Versus Pneumovax 23 Vaccine Response in the Diagnosis of Specific Polysaccharide Antibody Deficiency
Brief Title: Polysaccharide Antibody Response Study
Acronym: PARS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S57605
Record Dates: First submitted 2015-02-19; First posted 2015-04-29 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Specific Polysaccharide Antibody Deficiency
Keywords: Pneumovax 23; Typhim Vi; allohemagglutinins
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy controls (Experimental): Healthy volunteers who consented to participate in the study will be immunized with both Pneumovax 23 and Typhim Vi .
  Interventions: Biological: Pneumovax 23 (Sanofi Pasteur MSD); Biological: Typhim Vi (Sanofi Pasteur MSD)
- Patients (Experimental): Patients presenting for immune evaluation because of recurrent ENT/lung infection or invasive infection with encapsulated bacteria, in whom evaluation of pneumococcal antibody response is indicated, will be immunized with both Pneumovax 23 and Typhim Vi .
  Interventions: Biological: Pneumovax 23 (Sanofi Pasteur MSD); Biological: Typhim Vi (Sanofi Pasteur MSD)

INTERVENTIONS:
Biological: Pneumovax 23 (Sanofi Pasteur MSD) — Intramuscular injection of Pneumovax 23 vaccine (0.5 ml).
Biological: Typhim Vi (Sanofi Pasteur MSD) — Intramuscular injection of Typhim Vi vaccine (0.5 ml).

SUMMARY:
Specific polysaccharide antibody deficiency (SPAD) is a primary immunodeficiency characterized by a deficient antibody production to capsular polysaccharides with normal total immunoglobulin levels. Patients suffer from recurrent ear-nose and throat infections and lung infections. SPAD can also occur as part of a primary immunodeficiency affecting other components of the immune system. Diagnosis of SPAD is hampered by difficulties with the interpretation of the Pneumovax 23 antibody response. The purpose of this study is to assess the diagnostic value of the Typhim Vi antibody response and allohemagglutinin titers as an alternative to the Pneumovax 23 response to detect polysaccharide specific antibody deficiency.

DETAILED DESCRIPTION:
Healthy controls (n = 100) and patients with suspected SPAD (n = 100) will be immunized with both Pneumovax 23 and Typhim Vi (age 18 months - 55 years). Analyses of anti-pneumococcal polysaccharide antibodies and anti-Vi antibodies are performed before and 3-4 weeks after vaccination. Also bloodgroup and anti-A/anti-B are assessed. Relevant clinical information (ENT infections, lung infections, bronchiectasis, invasive infections) is obtained from the patient file and history and is noted in a Case Report Form.

The diagnostic performance of Typhim Vi response and allohemagglutinins will be analyzed by calculating sensitivity, specificity, predictive values, likelihood ratios and Receiver Operating Characteristic curves for Typhim Vi and allohemagglutinins using pneumococcal antibody response as the reference standard. The association between low Typhim Vi response or low allohemagglutinins and clinical signs of polysaccharide antibody deficiency will be studied by multiple logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Assessment of polysaccharide antibody response is indicated for the clinical care of the patient (not for healthy volunteers)
* Informed consent given

Exclusion Criteria:

* History of serious adverse reaction to a vaccine
* Vaccination with Typhim Vi or Pneumovax 23 in 5 years prior to the study
* (Potential) pregnancy

Ages: 18 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Typhim Vi response specific anti-Vi IgG as measured by ELISA | 3-4 weeks
  specific anti-Vi IgG as measured by ELISA
Pneumovax 23 response specific pneumococcal polysaccharide IgG as measured by ELISA | 3-4 weeks
  specific pneumococcal polysaccharide IgG as measured by ELISA

SECONDARY OUTCOMES:
allohemaglutinin titer as measured by column agglutination | 1 day
  bloodgroup, anti-A, anti-B IgG and IgM as measured by column agglutination
ENT infections (number of ENT infections obtained by history and medical file) | 12 months before inclusion untill inclusion
  number of ENT infections obtained by history and medical file
pneumonia (number of lung infections, confirmed on chest radiography, obtained by history and medical file) | 5 years before inclusion untill inclusion
  number of lung infections, confirmed on chest radiography, obtained by history and medical file
invasive infections (number and infection site of invasive infections obtained by history and medical file) | 5 years before inclusion untill inclusion
  number and infection site of invasive infections obtained by history and medical file
bronchiectasis (presence or absence of bronchiectasis (diagnosed by high resolution CT) obtained by history and medical file) | 5 years before inclusion untill inclusion
  presence or absence of bronchiectasis (diagnosed by high resolution CT) obtained by history and medical file
adverse effects | 4 weeks
  vaccine related adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Meyts, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Schaballie H, Vermeulen F, Verbinnen B, Frans G, Vermeulen E, Proesmans M, De Vreese K, Emonds MP, De Boeck K, Moens L, Picard C, Bossuyt X, Meyts I. Value of allohaemagglutinins in the diagnosis of a polysaccharide antibody deficiency. Clin Exp Immunol. 2015 May;180(2):271-9. doi: 10.1111/cei.12571. PMID 25516411